CLINICAL TRIAL: NCT04926870
Title: Application of CBL Teaching Based on PACS System in Training of Ophthalmologists
Brief Title: PACS System in the Training of Ophthalmologists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huijing Ye, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2021ye
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Case Based Learning
Keywords: teaching effect; teaching method
MeSH Terms: interventions — Radiology Information Systems

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PACS group (Experimental): PACS administration during teaching
  Interventions: Other: picture archiving and communication system
- Traditional group (Active Comparator): Traditional teaching without PACS
  Interventions: Other: traditional

INTERVENTIONS:
Other: picture archiving and communication system — PACS administration during teaching
  Other Names: PACS
  Arms: PACS group
Other: traditional — Clinical experience administration during teaching without PACS
  Other Names: Clinical experience teaching
  Arms: Traditional group

SUMMARY:
The purpose of this study is to evaluate teaching effect of CBL (case based learning) teaching method based on PACS (picture archiving and communication systems).

DETAILED DESCRIPTION:
In this randomized controlled clinical trial, we aim to explore the teaching effect of CBL (case based learning) teaching method based on PACS (picture archiving and communication systems) for doctors to master the specialized knowledge of orbital tumor.

ELIGIBILITY:
Inclusion Criteria:

* Orbital diseases standardized training of doctors
* Willing to receive training

Exclusion Criteria:

* Refuse to attend the assessment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Examination score | 3 months
  Examination score after training, with higher scores mean a better outcome. The highest score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Huijing, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China